CLINICAL TRIAL: NCT04593030
Title: Replication of the ARISTOTLE Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-ARISTOTLE
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Apixaban: Exposure group
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Warfarin — Warfarin dispensing claim is used as the reference
  Groups: Warfarin
Drug: Apixaban — Apixaban dispensing claim is used as the exposure
  Groups: Apixaban

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates: Market availability of apixaban in the U.S. started on December 28, 1012. For Marketscan: Jan 1, 2013 -Dec 31, 2018 (end of data availability). For Optum: Jan 1, 2013-Dec 31, 2019 (end of data availability). For Medicare: Jan 1, 2013 -Dec 31, 2017.

Inclusion Criteria:

* 1. Age ≥ 18 years
* 2. Atrial fibrillation - either of the following:

  * 2a. In atrial fibrillation or atrial flutter not due to a reversible cause and documented by ECG at the time of enrollment
  * 2b. If not in atrial fibrillation/flutter at the time of enrollment, must have atrial fibrillation/flutter documented on two separate occasions, not due to a reversible cause at least 2 weeks apart in the 12 months prior to enrollment. Atrial fibrillation/flutter may be documented by ECG, or as an episode lasting at least one minute on a rhythm strip, Holter recording, or intracardiac electrogram (from an implanted pacemaker or defibrillator)
* 3. One or more of the following risk factor(s) for stroke:

  * 3a. Age 75 years or older
  * 3b. Prior stroke, TIA, or systemic embolus
  * 3c. Either symptomatic congestive heart failure within 3 months or left ventricular dysfunction with an LV ejection fraction (LVEF) ≤ 40% by echocardiography, radionuclide study or contrast angiography
  * 3d. Diabetes mellitus
  * 3e. Hypertension requiring pharmacological treatment

Exclusion Criteria:

* 2. Clinically significant (moderate or severe) mitral stenosis
* 3. Increased bleeding risk that is believed to be a contraindication to oral anticoagulation (e.g. previous intracranial hemorrhage)
* 4. Conditions other than atrial fibrillation that require chronic anticoagulation (e.g. prosthetic mechanical heart valve)
* 5. Persistent, uncontrolled hypertension (systolic BP > 180 mm Hg, or diastolic BP > 100 mm Hg)
* 6. Active infective endocarditis
* 11. Simultaneous treatment with both aspirin and a thienopyridine (e.g., clopidogrel, ticlopidine)
* 12. Severe comorbid condition with life expectancy of ≤ 1 year
* 13. Active alcohol or drug abuse, or psychosocial reasons that make study participation impractical
* 14. Recent ischemic stroke (within 7 days)
* 15. Severe renal insufficiency (serum creatinine > 2.5 mg/dL or a calculated creatinine clearance < 25 mL/min, See Section 6.3.2.2)
* 17. Platelet count ≤ 100,000/ mm3
* 18. Hemoglobin < 9 g/dL
* 19. Women of child bearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing apixaban to warfarin. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of apixaban or the comparator drug (cohort entry date). Follow-up for the outcome, begins the day after drug initiation.
Sampling Method: Probability Sample
Enrollment: 220518 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke and Systemic Embolism | [Time Frame: Through study completion (a median of 98 days)]
  Relative hazard of composite outcome of Stroke and Systemic Embolism - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Franklin, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04593030/Prot_SAP_001.pdf